CLINICAL TRIAL: NCT02311712
Title: Non-endoscopic Esophageal Cancer Screening Program in Northern Iran
Brief Title: Non-endoscopic EC Screening Program in Northern Iran
Acronym: NESP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Waiting to receive capsule sponge device from the manufacturer.
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: International Agency for Research on Cancer (Other); University of Cambridge (Other); Golestan University of Medical sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 93-03-37-27139
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Early detection; Cytological examination
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (2):
- Capsule sponge (Active Comparator): Capsule sponge cytology examination coupled with H&E staining analysed for the presence of atypia and p53 immunohistochemistry
  Interventions: Device: Capsule sponge
- Control (No Intervention): No intervention

INTERVENTIONS:
Device: Capsule sponge — Capsule sponge cytology examination coupled with H&E staining analysed for the presence of atypia and p53 immunohistochemistry
  Arms: Capsule sponge

SUMMARY:
The aim of this study is to assess the effects of implementation of a non-endoscopic esophageal cancer-screening program on outcomes of interest in an asymptomatic high-risk population in Golestan Province, Iran. Study population will be recruited in two arms. In the intervention arm, cytological examination of the esophagus will be performed using a capsule sponge device. Subjects in the control arm will receive no intervention. All participants will be followed for 5 years. The outcomes of interest, including the incidence of esophageal cancer as well as mortality rates, will be compared between the two groups.

DETAILED DESCRIPTION:
Background:

Esophageal cancer (EC) is the 8th most common cancer and the 6th most common cause of death from cancer worldwide. Golestan province located in Northern Iran has been known as a high-risk area for esophageal squamous cell carcinoma (ESCC). Recent reports suggest an increasing rate of esophageal adenocarcinoma (EAC) in this region as well. Designing and implementing of screening programs may be effective for controlling these cancers. The investigators aim to develop a screening program for esophageal cancer in this region. The pilot phase of this project, the Golestan EC Screening Program (GESP), was conducted during 2011 and 2012 among 300 asymptomatic participants of Golestan Cohort Study (GCS), which is a prospective population-based cohort of 50,045 individuals, aged 40-75 years at baseline, in the eastern half of Golestan Province, Iran. The initial results of the GESP project showed a low participation rate for endoscopic screening. In other words, endoscopic ESCC screening was not feasible in our population, suggesting the need for a non-endoscopic screening method. Further results of the GESP project suggested that capsule sponge cytology is a feasible and valid primary method for ESCC screening in this region. Because of the promising findings of the GESP project, it has been decided to start the main phase of the EC screening program, called the "Non-endoscopic EC Screening Program in Northern Iran (NESP)". The aim of this study is to assess the effects of implementation of a non-endoscopic EC screening program on outcomes of interest in an asymptomatic high-risk population in Golestan Province, Iran.

Methods:

For sample size calculations, the investigators considered different scenarios based on the published literature and unpublished data. The prevalence of high grade dysplasia in the general population of Golestan has been estimated to be 1.4-3.6%. The sensitivity of cytological detection of esophageal squamous dysplasia (ESD) was predicted to be about 46% based on studies from China, and 60-100% based on studies from Iran, and according to previous studies, 27-65% of ESD lesions progress to invasive ESCC without treatment. The investigators used a rather conservative assumption to calculate sample size: a dysplasia prevalence of 1.5%, a 60% sensitivity for the sponge cytology, and a 2% progression to invasive ESCC in the screened (and treated) group vs. 40% in the untreated group. The investigators also assumed a power of 90%, a mean cluster size of 28 based on the PolyIran study (CV=0.84%), and an intra-class correlation (ICC) of 0.01. Based on these assumptions the investigators will need 4980 people in each arm. So, the investigators need to enroll 9,960 GCS participants > 50 years old. Estimating a 20% lack of consent, the final invitation lists of NESP project will consist of 12000 GCS participants including 6000 subjects in the intervention (capsule sponge) arm and 6000 subjects in the control arm.

A list of 12000 subjects from GCS participants will be prepared. Sampling will be done using a cluster randomization method. Each village will be considered as a cluster. Clusters will randomly be allocated into two groups, the intervention group (group 1) and the control group (group 2). Capsule sponge examination will be performed for all subjects in intervention clusters. But, participants in control clusters will be enrolled without capsule sponge examination. Both intervention and control subjects will be offered endoscopy if they develop upper GI symptoms according to current clinical practice.

The process of data collection and sampling will be performed at the community level. The NESP enrollment team will go to healthcare houses located in each village and data collection and sampling will be done there.

After obtaining informed consent, a structured questionnaire including data on demographic, socioeconomic status and medical history will be completed for each subject. Subjects will also be asked to fill in a quality of life (QOL) questionnaire. The investigators will use the validated Persian version of the WHOQOL-BREF questionnaire which was basically developed by the World Health Organization (WHO).

Then the capsule sponge examination will be performed for each subject in the community clinic after an overnight fast. The cytological specimen will be placed in preservative fluid and transferred to the histopathology lab.

Cytological specimens will be processed into paraffin blocks, and slides will be prepared from each paraffin block and will be stained using the hematoxylin and eosin (H&E) method. Cytological examination of the capsule sponge H&E slides will be done by expert pathologists.

The result will be reported according to the Bethesda system. All subjects with cytological diagnosis of atypia will be referred to "ATRAK clinic" (a central clinic for upper gastrointestinal disease in GONBAD, Iran) for endoscopic examination. Endoscopic examination with Lugol's iodine staining will be performed by previously described methods and biopsies will be taken from abnormal lesions. Histological examination of endoscopic biopsy samples will be done by expert pathologists. If the results of the endoscopic examination show high-grade dysplasia or cancer, the subject will be referred for treatment. These subjects will be treated with endoscopic mucosal resection (EMR) and/or radiofrequency ablation (RFA).

Participants will be followed annually according to the protocol of the GCS follow-up. Each subject will annually be contacted by a telephone call, and questions about the subject's vital status and cancer incidence will be asked from the subject or a first-degree relative. In addition, official data on subject's vital status will be obtained from the death registry unit in the Department of Health of Golestan University of Medical Sciences. Data on cancer incidence in the study subjects will also be obtained from the Golestan population-based cancer registry.

Both groups will be followed for 5 years. At the end of the study, the QOL questionnaire will be completed again for all available subjects.

The risk of developing outcomes will be compared between the intervention and control groups. Odds ratios and 95% confidence intervals (CI) will be calculated. Survival analysis will be done to assess survival rates in the sponge and control groups. The log rank test will be used to compare the survival rates between the two groups. Hazard ratios and 95% CI will be calculated for different variables using Cox regression analysis. Changes in QOL scores during the 5 year follow-up period will be compared between the sponge and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants of Golestan Cohort study with age higher than 50 years.

Exclusion Criteria:

* Subjects with a history of malignant disease, liver cirrhosis, or chronic renal failure will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Histologically-confirmed esophageal squamous cell carcinoma | 5 years
  Number of participants with Histologically-confirmed esophageal squamous cell carcinoma will be identified in both intervention and control arms
Death from Esophageal Squamous Cell Carcinoma | 5 years
  Number of Death from Esophageal Squamous Cell Carcinoma will be identified in both intervention and control arms
Death from all causes | 5 years
  Number of Death from all causes will be identified in both intervention and control arms

SECONDARY OUTCOMES:
Histologically-confirmed esophageal adenocarcinoma | 5 years
  Number of participants with Histologically-confirmed esophageal adenocarcinoma will be identified in both intervention and control arms
Histologically-confirmed gastric cardia adenocarcinoma | 5 years
  Number of participants with Histologically-confirmed gastric cardia adenocarcinoma will be identified in both intervention and control arms
Change in Quality of life | 5 years
  Change in Quality of life will be identified in both intervention and control arms

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, MD, Principal Investigator — Tehran University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Ervik M, Dikshit R, Eser S, Mathers C, et al. GLOBOCAN 2012 v1.0, Cancer Incidence and Mortality Worldwide: IARC CancerBase No. 11. Lyon, France: International Agency for Research on Cancer; 2013.
- [Background] Mahboubi E, Kmet J, Cook PJ, Day NE, Ghadirian P, Salmasizadeh S. Oesophageal cancer studies in the Caspian Littoral of Iran: the Caspian cancer registry. Br J Cancer. 1973 Sep;28(3):197-214. doi: 10.1038/bjc.1973.138. PMID 4743904
- [Background] Ghasemi-Kebria F, Roshandel G, Semnani S, Shakeri R, Khoshnia M, Naeimi-Tabiei M, Merat S, Malekzadeh R. Marked increase in the incidence rate of esophageal adenocarcinoma in a high-risk area for esophageal cancer. Arch Iran Med. 2013 Jun;16(6):320-3. PMID 23725063
- [Background] Roshandel G, Khoshnia M, Sotoudeh M, Merat S, Etemadi A, Nickmanesh A, Norouzi A, Pourshams A, Poustchi H, Semnani S, Ghasemi-Kebria F, Noorbakhsh R, Abnet C, Dawsey SM, Malekzadeh R. Endoscopic screening for precancerous lesions of the esophagus in a high risk area in Northern Iran. Arch Iran Med. 2014 Apr;17(4):246-52. PMID 24724600
- [Background] Etemadi A, Abnet CC, Golozar A, Malekzadeh R, Dawsey SM. Modeling the risk of esophageal squamous cell carcinoma and squamous dysplasia in a high risk area in Iran. Arch Iran Med. 2012 Jan;15(1):18-21. PMID 22208438
- [Background] Pan QJ, Roth MJ, Guo HQ, Kochman ML, Wang GQ, Henry M, Wei WQ, Giffen CA, Lu N, Abnet CC, Hao CQ, Taylor PR, Qiao YL, Dawsey SM. Cytologic detection of esophageal squamous cell carcinoma and its precursor lesions using balloon samplers and liquid-based cytology in asymptomatic adults in Llinxian, China. Acta Cytol. 2008 Jan-Feb;52(1):14-23. doi: 10.1159/000325430. PMID 18323271
- [Background] Taylor PR, Abnet CC, Dawsey SM. Squamous dysplasia--the precursor lesion for esophageal squamous cell carcinoma. Cancer Epidemiol Biomarkers Prev. 2013 Apr;22(4):540-52. doi: 10.1158/1055-9965.EPI-12-1347. PMID 23549398
- [Background] Solomon D, Davey D, Kurman R, Moriarty A, O'Connor D, Prey M, Raab S, Sherman M, Wilbur D, Wright T Jr, Young N; Forum Group Members; Bethesda 2001 Workshop. The 2001 Bethesda System: terminology for reporting results of cervical cytology. JAMA. 2002 Apr 24;287(16):2114-9. doi: 10.1001/jama.287.16.2114. PMID 11966386
- [Background] Roshandel G, Sadjadi A, Aarabi M, Keshtkar A, Sedaghat SM, Nouraie SM, Semnani S, Malekzadeh R. Cancer incidence in Golestan Province: report of an ongoing population-based cancer registry in Iran between 2004 and 2008. Arch Iran Med. 2012 Apr;15(4):196-200. PMID 22424034
- [Background] Roshandel G, Merat S, Sotoudeh M, Khoshnia M, Poustchi H, Lao-Sirieix P, Malhotra S, O'Donovan M, Etemadi A, Nickmanesh A, Pourshams A, Norouzi A, Debiram I, Semnani S, Abnet CC, Dawsey SM, Fitzgerald RC, Malekzadeh R. Pilot study of cytological testing for oesophageal squamous cell dysplasia in a high-risk area in Northern Iran. Br J Cancer. 2014 Dec 9;111(12):2235-41. doi: 10.1038/bjc.2014.506. Epub 2014 Sep 23. PMID 25247319